CLINICAL TRIAL: NCT06374537
Title: Evaluating the Impact of Targeted Physical Activity on Clinically Debilitated Dialysis Patients.
Brief Title: Evaluate the Impact of Targeted Physical Activity on Clinically Debilitated Dialysis Patients.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Enrico Benedetti, MD, Professor and Head Department of Surgery, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0784
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Frailty; Pain, Chronic; Dialysis; Complications; Kidney Diseases
MeSH Terms: conditions — Frailty; Chronic Pain; Kidney Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigate the effects of an exercise intervention on clinically debilitated dialysis patients. (Experimental): 150 patients from UI Health (≥ 18 years of age), who are on dialysis, or have chronic kidney disease stage 4 (CKD 4 = GFR between 15 and 29), or have chronic kidney disease stage 5 (CKD 5 = GFR below 15) and are considered clinically debilitated by their direct healthcare professional. After the initial baseline visit, subjects will come twice weekly, for roughly 1 hour each session, for 12 months (96 visits total). Subjects will also come in for data collection visits at baseline (prior to starting the exercise program), 6 months, and 12 months. Each of those visits will take about 2-3 hours. All testing done in the 3 test visits will help assess the patient's cardiovascular and functional responses and/or changes to the exercise intervention.
  Interventions: Other: Muscle Therapy
- Control (No Intervention): The control arm will receive no exercise intervention. Subjects will also come in for data collection visits at baseline (prior to starting the exercise program), 6 months, and 12 months. Each of those visits will take about 2-3 hours. All testing done in the 3 test visits will help assess the patient's cardiovascular and functional responses.

INTERVENTIONS:
Other: Muscle Therapy — Participants will attend 2 muscle therapy sessions a week for 12 months, for one hour each.
  Other Names: Targeted physical activity, Exercise
  Arms: Investigate the effects of an exercise intervention on clinically debilitated dialysis patients.

SUMMARY:
This research is being done to better understand the impact of the use of a specific physical activity training program (GH Method) in dialysis/kidney disease patients.

DETAILED DESCRIPTION:
The 12-Month Randomized Trial Group will include a total of 150 patients from UI Health (≥ 18 years of age), who are on dialysis, or have chronic kidney disease stage 4 (CKD 4 = GFR between 15 and 29) or have chronic kidney disease stage 5 (CKD 5 = GFR below 15) and are considered clinically debilitated by their direct healthcare professional will be enrolled. Randomization will be a 2:1 ratio (100 intervention, 50 control). The intervention arm will perform a 12-month exercise intervention which involves two days a week of personalized exercise rehabilitation. The control arm will receive no exercise intervention. Both arms of patients will be tested on various measures of health and function both at baseline (prior to intervention) at 6 months, and at 12 months (post intervention). This study will also investigate the effects of an exercise intervention on a subgroup of pre- and post- kidney transplant patients (PPKT Subgroup). This subgroup will include a total of 100 patients (≥ 18 years of age), who are on dialysis, or have CKD stage 4 or 5, and are considered clinically debilitated by their direct healthcare professional will be enrolled, or post- renal (kidney) transplant. This subgroup will perform 36 visits of exercise intervention which involves two days a week of personalized exercise rehabilitation. The Investigator will also utilize validated surveys and assessment tools to assess health issue management and depression severity.

ELIGIBILITY:
Inclusion Criteria:

* Clinically debilitated patients, currently on dialysis, or have CKD 4 (GFR between 15 and 29), or have CKD 5 (GFR below 15), or post- kidney transplant (for PPKT Subgroup only) as stated by patient's health care professional.
* Adequate cognitive ability to complete the questionnaires, give consent for the study and follow the physical and diet instructions

Exclusion Criteria:

* cardiac/pulmonary disease that contraindicate the physical training
* Unable to give consent
* Unable to travel to the training center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-05-22 (Actual); Primary Completion 2026-05-22 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Rate at which subjects will see changes in their physical abilities. | 12 months
  Participants will see improvements in their physical abilities after 12 months in the exercise training sessions. This will be assessed by comparing baseline, 6 months, 12 months, using a Short Physical Performance Battery test. This test requires the assessment of walking speed (time to walk 3 meters), a balance test (standing in 3 different positions for 10 seconds each-tandem, semi tandem, and side by side), and the time it takes to sit and stand 5 times in a chair (see above). Scoring is based on a scale of 0-12, lower numbers representing worse performance.

SECONDARY OUTCOMES:
Rate at which exercise will change body composition | 12 months
  With this hypothesis the Investigator will test whether muscle mass (DEXA scan) changes after 6 months and 12 months of an exercise intervention. Baseline measurement will be performed before the intervention, at 6 months and 12 months , with muscle mass measured by DEXA.
Rate at which exercise will change handgrip strength. | 12 months
  With this hypothesis the Investigator will test whether muscle strength (dynamometer) changes after 6 months and 12 months of an exercise intervention. Baseline measurement will be performed before the intervention, at 6 months and 12 months, with strength measured by dynamometer.
Rate at which subjects enrolled in the exercise intervention will have an overall changed sense of well-being. | 12 months
  Participants will be asked about their overall general health using the PROMIS.
Rate at which subjects enrolled in the exercise intervention will have an overall changed in their quality of life. | 12 months
  Participants will be asked about their mental health using SF 36.
Rate at which subjects enrolled in the exercise intervention will have an overall decreased change in depression. | 12 months
  Participants will be asked about their mental health using the BDI.
Rate at which subjects enrolled in the exercise intervention will have an overall change in pain intensity. | 12 months
  Participants will be asked about their overall pain intensity using the Numeric Rating Scale for Pain.

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Benedetti, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/37/NCT06374537/Prot_SAP_000.pdf